CLINICAL TRIAL: NCT04746742
Title: Tunneled Femoral Catheter Versus Femoro-femoral Arteriovenous Graft as a Lower-Extremity Hemodialysis Vascular Access: A Randomized Controlled Trial
Brief Title: Prosthetic Femoral Access for Haemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed Mosallam Mohammed Ibrahim, Specialist of Vascular Surgery, MD candidate, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MD.20.11.387
Record Dates: First submitted 2021-01-10; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Vascular Access Complication
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tunneled femoral catheter (Active Comparator): 20 patients with end stage renal disease and exhausted upper-extremity and chest-wall vascular accesses will be randomly allocated to this group
  Interventions: Procedure: Tunneled Femoral Catheter (TFC) group
- Femoral artery-femoral arteriovenous graft (Active Comparator): a straight or loop configuration 28patients with end stage renal disease and exhausted upper-extremity and chest-wall vascular accesses will be randomly allocated to this group
  Interventions: Procedure: Femoro-femoral Arteriovenous graft (FF-AVG) group

INTERVENTIONS:
Procedure: Tunneled Femoral Catheter (TFC) group — Patients with end-stage chronic kidney disease exhausted upper-extremity and chest-wall vascular accesses will be submitted to creation of a Lower-Extremity Hemodialysis Vascular either through application of tunneled femoral catheter
  Arms: Tunneled femoral catheter
Procedure: Femoro-femoral Arteriovenous graft (FF-AVG) group — Patients with end-stage chronic kidney disease exhausted upper-extremity and chest-wall vascular accesses will be submitted to creation of a Lower-Extremity Hemodialysis Vascular either through application of tunneled femoral catheter
  Arms: Femoral artery-femoral arteriovenous graft

SUMMARY:
This study will compare the outcomes of tunneled femoral catheter and femoro-femoral arteriovenous graft as a bailout procedure for hemodialysis in chronic kidney disease patients with exhausted upper-extremity and chest-wall vascular accesses regarding survival rate, complications, and quality of life

DETAILED DESCRIPTION:
Aim of the Work:

The aim of this work is to compare the outcomes of tunneled femoral catheter (TFC) and femoro-femoral AVG as regards survival, complication and quality of life as bailout procedure for hemodialysis in CRF patient with exhausted upper limb extremity and chest wall vascular accesses.

Patients and Methods:

Study Design and setting:

This is a single-centre prospective randomized controlled trial that will be conducted in The Vascular Surgery Department, Mansoura University Hospital, during the period from November 2020 to November 2022. It will be submitted for approval by Institutional Review Board, faculty of medicine, Mansoura University.

Eligibility criteria:

The study population will be on patients referred to the vascular surgery department suffering from end-stage renal disease (ESRD) with exhausted upper-extremity and chest wall vascular accesses.

Inclusion:

In this study, The investigator will include all ESRD patients belonging to the age group (≥ 15 years) who complain of exhaustion of all upper extremity vascular accesses.

Exclusion:

The investigators will exclude patients with previous history or evident deep venous thrombosis (DVT), varicose veins, femoral vein stenosis, arterial insufficiency, severe groin or limb infection.

Preoperative assessment:

A comprehensive history will be taken from the patients with regard to patient's demographics, underlying medical conditions, duration since the starting of haemodialysis, previous trials of vascular access, history of DVT and arterial insufficiency.

Also, patients will be examined to exclude any possibility for upper extremity vascular access. A meticulous examination of both lower limbs is done to assess the possibility of infection, signs of venous stenosis or arterial inefficiency including palpation of accessible lower limb arteries.

Routine laboratory investigations are carried out for all patients including complete blood count, liver function tests, renal function tests, arterial blood gases, bleeding and coagulation profiles, fasting and 2hr-postprandial serum glucose level, lipid profile, and glycosylated hemoglobin (HbA1c).

Further investigations include duplex ultrasonography (US) assessing for both superficial and deep venous system of the both lower limb. Bilateral lower limb arterial duplex is done to exclude any arterial disease. Also, a preoperative venous mapping of lower limb veins is mandatory.

Procedures and Postoperative care:

Procedures:

1. Tunneled femoral catheter: a standard technique is adopted according to the study performed by Herzallah using long tunneled catheter.
2. Femoral artery-femoral arteriovenous graft: a straight or loop configuration Ponikvar

Endpoints and Follow-up:

Every patient will be followed every week until first month, then every 3 months until the end of the first years so that the hemodynamic improvement will be assessed.

Primary outcome:

• Evaluation of primary patency rates within the study follow-up time frame.

* In case of TFC: Normally an extracorporeal blood flow should be about 300 ml/min. based on this, the catheter dysfunction can be defined by the first occurrence of either peak blood flow of 200 ml per minute or less for 30 minutes during a dialysis treatment, mean blood flow of 250 ml per minute or less during two consecutive dialysis treatments, or inability to initiate dialysis owing to inadequate blood flow, after attempts to restore patency have been attempted.
* In case of AVG, stenosis > 50% of the prosthesis diameter or complete occlusion is considered significant. This can be assessed by duplex ultrasonography every six months or when the patency is questionable.

The patency rates will be determined according to the reporting standards, set by the Committee of Reporting Standards for arteriovenous hemodialysis accesses

Secondary outcome:

* The secondary patency: the patency rates will be determined according to the reporting standards, set by the Committee of Reporting Standards for arteriovenous hemodialysis accesses
* The special adverse events complicating lower-extremity hemodialysis access. The severity of arteriovenous access complications will be graded according to the Reporting Standards document . Complications are defined according Clavien-Dindo.
* Patient satisfaction will be assessed using a validated tool, the vascular access score questionnaire, at 6 and 12 months postoperatively.
* Besides, operative time, hospital stay, and survival rate will be assessed.

Sample size calculation:

Based on the average of the primary outcome (primary patency), a previous study showed that the mean rate in AVGs at 6 months was 53%, while another study showed that the mean rate in TFC at six months was 14%.

Using sample size calculation software (www.clincalc.com), a minimum of 44 patients will be needed to achieve a study power of 80% with alpha set at 5%. Estimating a drop-out rate and loss to follow-up of 10%, a total of 48 patients will be ultimately included.

Random sequence generation and blinding:

Patients will be randomized to one of two groups; group I Tunneled femoral catheter and group II Femoral artery-femoral vein graft.

Randomization will be undertaken by the sealed envelope method using randomization software. Neither the operating surgeons nor the assessors during the follow-up will be aware about patients' participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* All end-stage renal disease patients who complain of exhaustion of all upper-extremity and chest-wall vascular accesses.
* ≥ 15 years

Exclusion Criteria:

* patients with previous history or evident deep venous thrombosis
* varicose veins
* femoral vein stenosis
* arterial insufficiency
* severe groin or limb infection.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 12 months postoperatively
  In case of TFC: Normally an extracorporeal blood flow should be about 300 ml/min. based on this, the catheter dysfunction can be defined by the first occurrence of either (1) peak blood flow of 200 ml per minute or less for 30 minutes during a dialysis treatment, (2) mean blood flow of 250 ml per minute or less during two consecutive dialysis treatments, or (3) inability to initiate dialysis owing to inadequate blood flow, after attempts to restore patency have been attempted.
  - In case of AVG, stenosis > 50% of the prosthesis diameter or complete occlusion is considered significant. This can be assessed by duplex ultrasonography every six months or when the patency is questionable. The patency rates will be determined according to the reporting standards, set by the Committee of Reporting Standards for arteriovenous hemodialysis accesses.

SECONDARY OUTCOMES:
Secondary patency | 24 months
  the patency rates will be determined according to the reporting standards, set by the Committee of Reporting Standards for arteriovenous hemodialysis accesses.
Special adverse events complicating lower-extremity haemodialysis access | 24 months
  The severity of arteriovenous access complications will be graded according to the Reporting Standards document. Complications are defined according Clavien-Dindo.
Patient satisfaction | 6 & 12 months postoperatively
  assessed using a validated tool, the vascular access score questionnaire

OTHER OUTCOMES:
Operation time | 24 months
  From skin incision until skin closure
Hospital stay | 24 months
  From surgery until leaving the hospital
Survival rate | 24 months
  Incidence of patient who survive

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed Mosallam Mohammed Ibrahim, Al Mansurah, Dakahleyya, Egypt